CLINICAL TRIAL: NCT03821025
Title: Treatment of Malignant Distal Biliary Obstruction - a Randomized Study
Brief Title: Self-expandable Metal Stents Versus Multiple Plastic Stents for Palliation of Biliary Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Marc Bernon, Senior consultant, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 661/2017
Record Dates: First submitted 2019-01-26; First posted 2019-01-29 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Bile Duct Obstruction, Extrahepatic; Cancer of the Pancreas; Cancer of the Bile Duct; Biliary Stricture
MeSH Terms: conditions — Cholestasis, Extrahepatic; Pancreatic Neoplasms; Bile Duct Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multiple Plastic Stents (Active Comparator): Patients will receive two 8.5Fr Platic biliary stents placed side by side across the biliary stricture.
  Interventions: Device: Biliary stent
- Self-expandable Metal Stents (Active Comparator): Patients will receive a fully covered Self-expandable Metal Stents (10mm) across the biliary stricture
  Interventions: Device: Biliary stent

INTERVENTIONS:
Device: Biliary stent — Palliation of malignant biliary obstruction

SUMMARY:
A randomised clinical trial to compare the clinical efficacy of multiple plastic stents to fully covered self expanding metal stents in the palliation of distal malignant biliary obstruction in patients with irresectable tumours.

ELIGIBILITY:
Inclusion Criteria:

* 18years of age or older
* informed consent obtained after oral and written information
* clinical data in accordance with a malignant bile duct obstruction
* imaging evidence: (ultrasonography (US), computed tomography (CT) or magnetic resonance imaging (MRI) shows signs of extrahepatic malignant common bile duct obstruction
* typical ERCP findings of a malignant common bile duct stenosis
* proximal margin of the bile duct stenosis ≥2 cm from the hepatic confluence
* bilirubin > 50 micromol/L
* radical surgery not deemed possible

Exclusion Criteria:

* patients with active hepatitis or other jaundice-causing hepatic diseases
* informed consent not obtained or patient unable to give informed consent
* patients with no understanding of English, Afrikaans or Xhosa where it is not possible to obtain informed consent
* metastasis with multiple significant intrahepatic stenosis causing blockage of one or more segments of the liver (liver metastasis otherwise not an exclusion criteria)
* the patient is a possible candidate for surgical resection
* suspicion of a non-malignant bile duct obstruction, e.g. stones or benign stenosis (should initiate further investigations)
* the proximal end of the stenosis is < 2 cm from the hepatic confluence
* previous BII or Roux-en-Y gastric reconstruction
* significant duodenal obstruction making ERCP difficult
* previous bile duct stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients without stent failure | 12 months
  Number of patients without Stent failure (jaundice) or death with a patent stent

SECONDARY OUTCOMES:
Overall survival | 12 months
  Number of patietns alive in each group at 12 months
Stent deployment failure | During procedure
  Number of patients in whom there was failure to deploy the assigned stent(s) after randomisation
Cost | 12 months
  The differance in treatment costs between the two groups, measured in USD

CONTACTS AND LOCATIONS:
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No